CLINICAL TRIAL: NCT05846997
Title: Use of INnovative and Micro-INvasive TEchniques for the Early Identification of Breast Cancer Patients Benefitting From Neo-adjuvant Therapy
Acronym: INTENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2018-10
Record Dates: First submitted 2023-03-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Liquid biopsy and imaging — Liquid biopsy and imaging

SUMMARY:
The purpose of the study is the identification of novel micro-invasive predictors of pathological complete response (pCR) during neo-adjuvant therapy

DETAILED DESCRIPTION:
This is a single arm prospective, monocentric, open, experimental pilot study. The response to NAC in breast cancer is extremely heterogeneous. The study and the identification of factors that can predict the response to treatment is therefore a priority, constituting a relevant "clinical unmet need".Modern molecular biology techniques as well as imaging diagnostics could be valuable tools for characterizing the response to NAC toward the definition of more personalized therapies.The prediction of therapy response after two cycle of chemotherapy rather than at the end of six cycles using non-invasive procedures will spare unwanted toxicity to the patients and resources to the Regional and National Health system. This study will also provide the patients, their familiar and all the stakeholders involved in the cure of Breast Cancer new important information regarding the management of breast cancer patients.This is a non-interventional study; therefore, the treatment will be as per physician choice according to the most appropriate therapeutic opportunities available for each patients' based on the type and stage of disease and the patients' performance status.Currently, the NAC regimens commonly used at CRO-Aviano for NAC are Epirubicine 90 mg/mq + Ciclophosphamide 600 mg/mq d1 q21 or q14 (EC)(dose dense) followed by weekly Paclitaxel 80 mg/mq for a total of 12 administrations. Occasionally, due to patients and tumor features only weekly Paclitaxel is used, and usually in this case up to 24 administrations may be given. Only in the case of HER2 positive BC trastuzumab 2 mg/kg is added to weekly Paclitaxel. Given the low response rate of hormone-based neoadjuvant therapy, only in rare cases (e.g. patients not amenable of surgery due to comorbidities), this approach is used.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histological Diagnosis of Infiltrating Breast Cancer.
3. The presence of measurable mammary lesions;
4. The presence of metabolically active mammary lesions;
5. Performance Status (Eastern Cooperative Oncology Group scale, ECOG) ≤ 1;
6. Compliance with periodic blood withdrawal;
7. Compliance with periodic PET/CT and RMN imaging;
8. Adequate clinical and laboratory test results for undertaking neoadjuvant chemotherapy and surgery;
9. Written informed consent.

Exclusion Criteria:

1. The presence of contraindications for the execution of RMN and PET-TC;
2. Presence of metastatic disease;
3. Pre-existing or concurrent tumors, except in situ carcinoma or basophilic carcinoma of the skin;
4. Uncontrolled active infections;
5. Insufficient patient compliance;
6. Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Histological Diagnosis of Infiltrating Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-02-24 (Estimated)

PRIMARY OUTCOMES:
Identification of novel micro-invasive predictors of pathological complete response (pCR) during neo-adjuvant therapy. | from start of therapy until first documented progression, assessed up to 12 months
  1. Determine if a PET SUV decrease ≥ 50% after two cycles of therapy respect to the basal value will predict the pCR predict the pCR of breast cancer patients treated with neo-adjuvant therapy;
Identification of novel micro-invasive predictors of pathological complete response (pCR) during neo-adjuvant therapy. | from start of therapy until first documented progression, assessed up to 12 months
  2. Determine if a cfDNA variation ≥ 25% of the basal value after two cycles of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy

SECONDARY OUTCOMES:
Determine if the basal number of CTC and/or its variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy; | from start of therapy until first documented progression, assessed up to 12 months
  Determine if the basal number of CTC and/or its variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy;
Determine if the basal SERS spectra and/or its variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy pCR of breast cancer patients treated with neo-adjuvant therapy; | from start of therapy until first documented progression, assessed up to 12 months
  Determine if the basal Metabolomics spectra and/or its variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy;
Determine if the basal SERS spectra and/or its variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy; | from start of therapy until first documented progression, assessed up to 12 months
  Determine if the basal SERS spectra and/or its variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy;
Determine if the basal Cytokines serum levels and/or their variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy; | from start of therapy until first documented progression, assessed up to 12 months
  Determine if the basal Cytokines serum levels and/or their variation after two cycle of therapy will predict the pCR of breast cancer patients treated with neo-adjuvant therapy;
Determine if a the basal Immune proficiency will predict the pCR of breast cancer patients treated with neo-adjuvant therapy; | from start of therapy until first documented progression, assessed up to 12 months
  Determine if a variation in T cell sub-populations will predict the pCR of breast cancer patients treated with neo-adjuvant therapy;
Evaluate over time Relapse Free Survival (RFS) and correlate with micro-invasive parameters from primary and/or secondary objectives. | from start of therapy until first documented relapse, assessed up to 12 months
  Evaluate over time Relapse Free Survival (RFS) and correlate with micro-invasive parameters from primary and/or secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Nicoloso, MD, Principal Investigator — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico, Aviano, Pordenone, Italy